CLINICAL TRIAL: NCT04630275
Title: Vitality-Obs; An Observational and Descriptive Cross-sectional Study of Gonadal Dysfunction in Male Long-term Survivors of Malignant Lymphoma
Brief Title: Gonadal Dysfunction in Male Long-term Survivors of Malignant Lymphoma; Vitality-Obs
Status: Completed | Type: Observational
Sponsor: Lars Møller Pedersen (Other)
Responsible Party: Sponsor-Investigator, Lars Møller Pedersen, Senior Consultant, Herlev Hospital
Organization: Herlev Hospital (Other)
Other Study IDs: Vitality1
Record Dates: First submitted 2020-07-27; First posted 2020-11-16 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Hypogonadism
Keywords: lymphoma; Diffuse Large B-Cell Lymphoma; Hodgkin; hypogonadism; testosterone; EORTC; Quality of life; Sexuality; Sexual health; Cancer; IIEF-5; Doxorubicin; anthracycline; Leydig cells; Hypothalamus; adriamycin
MeSH Terms: conditions — Hypogonadism; Lymphoma; Lymphoma, Large B-Cell, Diffuse; Sexuality; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study is an observational cross-sectional study which aims to investigate the relationship between treatment with chemotherapy and the development of low levels of testosterone in the blood in patients cured for aggressive lymphoma. We hypothesize that patients in turn will develop sexual dysfunction and poor quality of life because of this reduced level of testosterone. Cancer treatment is increasingly effective and the overall survival higher, which makes issues like sexuality and long-term quality of life more and more important to address in cured cancer patients. Patient sexuality and quality of life is measured by 3 questionnaires filled out once, and serum testosterone by a single blood sample. If serum testosterone is in the lower part of the normal reference interval, patients will be offered further hormonal evaluation by department of growth and reproduction at Copenhagen University Hospital. We hope to show that future follow up visits should include focus on sexuality and serum testosterone. Questionnaires and blood samples can be implemented easily and without great cost.

DETAILED DESCRIPTION:
Diffuse large B-cell lymphoma and Hodgkin Lymphoma are two aggressive lymphomas often treated with doxorubicin containing chemotherapy. Doxorubicin is an anthracycline and is known to be toxic to both Leydig Cells of the testes and hormone-producing cells of the hypothalamus. Therefore patients treated with this drug are at risk of developing hypogonadism. Standard follow-up programs do not include investigation of hormone levels. With this study we aim to investigate the extent of hypogonadisme in patients treated with anthracycline containing chemotherapy, to clarify whether it is relevant to include serum testosterone in standard follow-up programs.

Our Hypothesis:

Hypothesis 1: A significant proportion of long-term male survivors of HL and DLBCL have impaired QoL due to sexual dysfunction.

Hypothesis 2: A significant proportion of long-term male survivors of HL and DLBCL have reduced levels of testosterone.

Hypothesis 3: A significant relationship between QoL, sexual dysfunction and testosterone levels exists.

To clarify the extent of hypogonadisme a single blood test including s-total-testosterone will be drawn once, and levels below age adjusted reference levels will be classified as hypogonadisme. To assess patients sexuality and quality of life, 3 questionnaires will be filled out; the EORTC QLQ-C30 for general quality of life, EORTC SHQ-22 for sexual health and IIEF-5 for sexual function.

To evaluate whether normal reference levels are sufficient in the examination of lymphoma survivors, included men with serum testosterone in the lower part of the normal reference interval will be offered further hormonal evaluation at the department of growth and reproduction at Copenhagen University hospital. Blood test results will be evaluted by this research group.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years at follow-up
2. Male
3. Verified diagnosis of de novo DLBCL or classical HL diagnosed between April 2008 and April 2018 according to WHO classification.
4. Completed curative intent first line treatment with anthracycline-containing chemotherapy with or without consolidating radiotherapy, with disease in complete remission at EOT-PET/CT at least one year prior to inclusion.
5. Literate in Danish

Exclusion Criteria:

1. Concurrent low-grade lymphoma
2. Current or prior lymphoproliferative disease of the central nervous system (CNS)
3. Current or prior lymphoproliferative disease of the testes
4. Mental or physical conditions that are expected to prevent the necessary "compliance" and/or "adherence" in relation to the study procedures.
5. Treatment with second line chemotherapy or high dose therapy.
6. Current or prior anabolic steroid drug abuse

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Will be based on social security number
Study Population: A cohort of patients with Hodgkin Lyphoma or Diffuse Large B-Cell Lymphoma diagnosed during the period April 2008- April 2018 at the Departments of Hematology, Herlev Hospital, Copenhagen University Hospital and Zealand University Hospital, will be identified through The Danish Lymphoma registry (LyFo).
Sampling Method: Non-Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-04-24 (Actual); Study Completion 2023-04-24 (Actual)

PRIMARY OUTCOMES:
Serum-testosterone level | At inclusion
  The frequency of sexual dysfunction measured by serum-testosterone level below age adjusted reference levels, in patients with DLBCL or HL.

SECONDARY OUTCOMES:
Frequency of co-morbidity according to Cumulative Illness Rating Scale (CIRS) score | At inclusion
  The prevalence of CIRS score above 6
Frequency of Erectile Function according to International Index of Erectile Function (IIEF-5) | At inclusion
  The frequency of IIEF-5 scores below 22
Level of sexual dysfunction symptoms | At inclusion
  According to SHQ-22 symptom scores. High symptoms scores represents high level of symptoms.
Level of sexual function | At inclusion
  According to SHQ-22 function scores. High symptoms scores represents high level of functioning.
Level of Quality of life, functioning | At inclusion
  According to QLQ-C30 function scores. High function scores represents a high level of functioning.
Level of Quality of life, symptoms | At inclusion
  According to QLQ-C30 symptoms scores. High symptoms scores represents high level of symptoms.
Level of Quality of life, global health | At inclusion
  According to QLQ-C30 global health scores. High symptoms scores represents high level of global health.
serum sex hormone binding globulin (SHBG) | Through study completion, up to two years after incusion.
  The frequency of serum SHBG levels above the reference level
Serum Luteinizing hormone (LH) | Through study completion, up to two years after incusion.
  The frequency of serum LH levels above the reference level
Serum Inhibin B | Through study completion, up to two years after incusion.
  The frequency of serum Inhibin B levels below the reference level
Serum Follicle stimulating hormone (FSH) | through study completion, up to two years after inclusion
  The frequency of serum FSH levels above the reference level
Serum Estradiol | through study completion, up to two years after inclusion
  The frequency of serum estradiol levels above the reference level
Serum INSL-3 | through study completion, up to two years after inclusion
  The frequency of serum estradiol levels below the reference level
Serum hemoglobin | through study completion, up to two years after inclusion
  The frequency of serum hemoglobin levels above the reference level
Serum hematocrit | through study completion, up to two years after inclusion
  The frequency of serum hematocrit levels above the reference level
Serum free testosterone | through study completion, up to two years after inclusion
  The frequency of serum free testosterone levels above the reference level

CONTACTS AND LOCATIONS:
Locations (3):
- Denmark (3):
  - Copenhagen University Hospital, Copenhagen
  - Herlev University Hospital, Herlev
  - Zealand University Hospital, Roskilde